CLINICAL TRIAL: NCT06031935
Title: Yoga for Adolescent Anterior Knee Pain
Brief Title: Yoga for Adolescent Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004289
Record Dates: First submitted 2023-08-23; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Adolescent
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga study group (Experimental): This is the only arm of the study. The patients will be given yoga videos to do at home for 8 weeks as a treatment for anterior knee pain.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — The patients will receive links to two yoga videos. They will do each of these videos at home for 4 weeks.

SUMMARY:
Adolescent atraumatic anterior knee pain is a common yet cumbersome diagnosis that is currently managed with home exercises and physical therapy. The goal of this project is to present patients with an alternative treatment in the form of yoga available in an online video format. This new treatment, in the form of online yoga videos, may be more preferred for some patients and allow for higher compliance with home exercises aimed at treating anterior knee pain.

DETAILED DESCRIPTION:
Adolescent atraumatic anterior knee pain is a common yet cumbersome diagnosis that is currently managed with home exercises and physical therapy. The goal of this project is to test the compliance and efficacy of an alternative treatment in the form of yoga available in an online video format. This study will help further the treatment understanding of one of the most common patient clinical presentations, atraumatic anterior knee pain in adolescents. This is a cumbersome patient presentation that is frustrating for both the patient and treating team in that there is no concrete treatment algorithm that works for everyone. Online yoga videos may be more preferred for some patients and allow for higher compliance with home exercises aimed at treating anterior knee pain. With this study, the investigators hope to ensure that the yoga videos provide equal, or more, pain relief and flexibility at the completion of the program.

It is hypothesized that patients completing the yoga program will have equivalent or greater flexibility, compliance, and pain relief when compared with current treatment recommendations for anterior knee pain.

This study aims to assess the success of a video-based eight-week home yoga program at improving compliance, increasing flexibility and functionality of knee movements. Compliance will be tracked through recorded access to the specific YouTube videos hosted through the CTPO YouTube Channel. Anterior knee pain patients will be given a link to two yoga videos and will be asked to do them at home, or wherever convenient for 8 weeks, 3-4 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Children with non-structural anterior knee pain

Exclusion Criteria:

* Any intra-articular injuries
* No access to internet
* Non-english speaking

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient Flexibility | Baseline and 8 weeks
  Popliteal angle to test hamstring flexibility. On a scale of 0-90. A popliteal angle of 90 would mean very tight hamstrings. Prone heel to buttocks measurement will be taken to determine how close the patient can get their heel to buttocks. It will be measured in inches. A larger measurement means less flexibility. 0" is an ideal measurement.

SECONDARY OUTCOMES:
Number of views of yoga videos | Log will be recorded weekly for 8 weeks.
  Patient will keep a log of the number of times they do the videos, and we will use YouTube analytics to confirm the number of views.
International Knee Documentation Committee (pedi-IKDC) Survey Score | baseline, 8 weeks and 4 months
  Patient Reported Outcome survey. On a scale of 0-100. 100 means knee is fully functional.
Yoga video satisfaction survey | 8 weeks and 4 months
  Satisfaction questions as defined by study team on a scale of 0-5. To determine if the yoga videos were useful to the patients.
Patient-Reported Outcomes Measurement Information Systems (PROMIS) pain interference scale | baseline, 8 weeks and 4 months
  Measures the extent that pain is interfering with the patient's daily lifestyle. Pain is measured on a T-scale. 50 is the median. 20-55 is considered within the normal limits. 70+ is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Ellington, MD, Principal Investigator — University of Texas at Austin, Central Texas Pediatric Orthopedics
Locations (1):
- Central Texas Pediatric Orthopedics, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared outside of the study team.

REFERENCES:
- [Background] Galantino ML, Galbavy R, Quinn L. Therapeutic effects of yoga for children: a systematic review of the literature. Pediatr Phys Ther. 2008 Spring;20(1):66-80. doi: 10.1097/PEP.0b013e31815f1208. PMID 18300936
- [Background] Donohue B, Miller A, Beisecker M, Houser D, Valdez R, Tiller S, Taymar T. Effects of brief yoga exercises and motivational preparatory interventions in distance runners: results of a controlled trial. Br J Sports Med. 2006 Jan;40(1):60-3; discussion 60-3. doi: 10.1136/bjsm.2005.020024. PMID 16371493
- [Background] Hainsworth KR, Liu XC, Simpson PM, Swartz AM, Linneman N, Tran ST, Medrano GR, Mascarenhas B, Zhang L, Weisman SJ. A Pilot Study of Iyengar Yoga for Pediatric Obesity: Effects on Gait and Emotional Functioning. Children (Basel). 2018 Jul 4;5(7):92. doi: 10.3390/children5070092. PMID 29973555